CLINICAL TRIAL: NCT05487235
Title: A Phase Ib, Open-Label Study Evaluating the Safety, Pharmacokinetics, and Activity of GDC-1971 in Combination With Atezolizumab in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Activity of GDC-1971 in Combination With Atezolizumab in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO43712; 2021-006479-40 (EudraCT Number)
Record Dates: First submitted 2022-07-21; First posted 2022-08-04 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors; Metastatic Solid Tumors
MeSH Terms: interventions — atezolizumab; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose-finding Stage: GDC-1971 (Experimental): Participants will receive GDC-1971 tablet or capsule at assigned dose, orally once daily (QD) on Days 1-21 of each cycle, along with atezolizumab 1200 milligrams (mg) intravenous (IV) infusion once every 3 weeks (Q3W), until unacceptable toxicity or loss of clinical benefit. A subset of participants will participate in evaluations regarding tablet versus (vs) capsule formulations.
  Interventions: Drug: GDC-1971; Drug: Atezolizumab
- Expansion Stage: GDC-1971 (Experimental): Participants will receive GDC-1971 orally at the assigned dose QD on Days 1-21 of each cycle and atezolizumab 1200 mg IV on Day 1 of each cycle until unacceptable toxicity or loss of clinical benefit. A subset of participants will participate in evaluations regarding tablet vs capsule formulation, the effect of food and acid-reducing agents on GDC-1971.
  Interventions: Drug: GDC-1971; Drug: Atezolizumab; Drug: Omeprazole

INTERVENTIONS:
Drug: GDC-1971 — Capsule or tablet administered orally.
  Other Names: RO7517834, RLY-1971
Drug: Atezolizumab — Administered as IV infusion.
  Other Names: RO5541267
Drug: Omeprazole — Administered orally as tablet or capsule in the acid-reducing agent assessment.
  Arms: Expansion Stage: GDC-1971

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics (PK), and activity of GDC-1971 when administered in combination with atezolizumab in participants with locally advanced or metastatic solid tumors.

The study will have 2 stages- dose finding stage and expansion stage. In expansion stage participants with non-small cell lung cancer programmed death ligand -1 high (NSCLC PD L-1 high), NSCLC PD L-1 low, head and neck squamous cell carcinoma (HNSCC) PD L-1 positive, BRAF wild type (BRAF WT) melanoma and any locally advanced or metastatic solid tumors will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Has Eastern Cooperative Oncology Group(ECOG) Performance Status of 0 or 1
* Has Life expectancy >= 12 weeks
* Adequate organ function
* Measurable disease per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1).

Inclusion Criteria for Dose-Finding Stage:

* Histologically confirmed locally advanced or metastatic solid tumor that has progressed after at least one available standard therapy or for which approved standard therapy has proven to be ineffective or intolerable

Inclusion Criteria for Expansion Stage: NSCLC Cohort

* Histologically confirmed locally advanced or metastatic NSCLC
* Absence of epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK)
* PD- L1 positive
* No prior systemic therapy for locally advanced or metastatic NSCLC

Inclusion Criteria for Expansion Stage: HNSCC Cohort

* Histologically confirmed recurrent, or metastatic HNSCC
* PD-L1 positive
* No prior systemic therapy for recurrent or metastatic HNSCC

Inclusion Criteria for Expansion Stage: BRAF WT melanoma Cohort

* Histologically confirmed locally advanced or metastatic or unresectable locally advanced cutaneous BRAF WT melanoma or melanomas of unknown primary that are non-mucosal and non -uveal that has progressed on or after treatment that included anti PD1 or anti PD-L1 therapy

Inclusion Criteria for Expansion Stage: Other Advanced or Metastatic Solid Tumors Cohort

* Histologically confirmed locally advanced or metastatic solid tumor that has progressed after at least one available standard therapy or for which approved standard therapy has proven to be ineffective or intolerable, standard therapy is considered inappropriate, or an investigational agent is a recognized standard of care

Exclusion Criteria:

* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases.
* Has leptomeningeal disease or carcinomatous meningitis
* Has uncontrolled hypertension
* Has left ventricular ejection fraction < institutional lower limit of normal or < 50%
* Has clinically significant history of liver disease including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Has an active or history of autoimmune disease or immune deficiency including myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or multiple sclerosis. Participants with a history of autoimmune- related hypothyroidism on thyroid replacement hormone or with controlled Type I diabetes mellitus on a stable dose of an insulin regimen are eligible for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Up to approximately 2.5 years
Percentage of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to 30 days after final dose of study treatment (up approximately to 2.5 years)
Percentage of Participants With Clinically Significant Change from Baseline in Clinical Laboratory Test Results | Baseline up to 30 days after final dose of study treatment (up approximately to 2.5 years)
Percentage of Participants With Clinically Significant Change From Baseline in RR and QT Intervals as Measured by Electrocardiogram (ECG) | Baseline up to 30 days after final dose of study treatment (up approximately to 2.5 years)
Percentage of Participants Experiencing Dose Limiting Toxicities (DLTs) | From Day 1 to Day 21 of Cycle 1 of the dose finding stage
Plasma Concentration of GDC-1971 | Up to approximately 2.5 years

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve From Time 0 to 96 hours (AUC0-96 hr) Following GDC-1971 Capsule or Tablet Administration | Up to approximately 2.5 years
AUC From Time 0 to Infinity (AUCinf) Following GDC-1971 Capsule or Tablet Administration | Up to approximately 2.5 years
Cmax of GDC-1971 Following Capsule or Tablet Administration | Up to approximately 2.5 years
AUC 0-96 hr Following GDC-1971 Tablet Administration Under Fasted and Fed Conditions | Up to approximately 2.5 years
AUC inf Following GDC-1971 Tablet Administration Under Fasted and Fed Conditions | Up to approximately 2.5 years
Cmax of GDC-1971 Following Tablet Administration Under Fasted and Fed Conditions | Up to approximately 2.5 years
AUC 0-24 hr at Steady State Following GDC-1971 Tablet Administration and in Combination With Omeprazole | Up to approximately 2.5 years
Cmax at Steady State Following GDC-1971 Tablet Administration and in Combination With Omeprazole | Up to approximately 2.5 years
Objective Response Rate (ORR) | Up to approximately 2.5 years
Duration of Response (DOR) | Up to approximately 2.5 years
Progression Free Survival (PFS) | Up to approximately 2.5 years
PFS Rate | Month 6
Overall Survival (OS) Rate | Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- Argentina (3):
  - Sanatorio Allende, Córdoba
  - Fundacion CORI para la Investigacion y Prevencion del Cancer, La Rioja
  - Centro Medico IPAM, Rosario
- Australia (5):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Border Medical Oncology, Wodonga, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Austin Hospital, Heidelberg, Victoria
  - One Clinical Research Perth, Nedlands, Western Australia
- Brazil (8):
  - Liga Paranaense de Combate Ao Cancer - Hospital Erasto Gaertner, Curitiba, Pará
  - Hospital de Clinicas de Porto Alegre HCPA PPDS, Pôrto Alegre, Pará
  - ONCOSITE Centro de Pesquisa Clínica Em Oncologia, Ijuí, Rio Grande do Sul
  - Fundacao Pio XII Hospital de Cancer de Barretos, Barretos, São Paulo
  - Fundação Doutor Amaral Carvalho - Hospital Amaral, Jaú, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose Do Rio Preto Hospital de Base - PPDS, São José do Rio Preto, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Instituto Brasileiro de Controle Do Câncer IBCC, São Paulo
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Auckland City Hospital, Auckland, New Zealand
- South Korea (5):
  - Chungbuk National University Hospital, Cheongju-si
  - National Cancer Center, Goyang-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center - PPDS, Seoul

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing
Supporting Information: Study Protocol, SAP, CSR